CLINICAL TRIAL: NCT04377802
Title: Safe Return to Regular Clinical Operation After COVID-19 Pandemic; (Oncology Center, Prospective Cohort)
Brief Title: Safe Return to Regular Clinical Operation After COVID-19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Fahad Specialist Hospital Dammam (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KFSH-ONC-02
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19 | interventions — Molecular Diagnostic Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: molecular testing for virus RNA using RT-PCR — Serological testing will be performed using SARS-CoV-2 IgG assay kit (Abbott Diagnostics, US) to check for the immunity. The IgG serology test (200 individuals per run) will be done using ARCHITECT i2000SR system which provides the results within 60 minutes

SUMMARY:
. Coronavirus (SARS-CoV2) appeared first in China late 2019 and caused an acute respiratory disease referred to as Coronavirus disease 2019 (COVID-19). SARS-CoV2 is considered by the World Health Organization (WHO) as pandemic and affected nations worldwide, leading to close borders and major economical struggle. The ongoing viral threat due to the lack of effective therapies and vaccination might prolonged this economical challenge and many businesses will face huge financial constraints leading to laying off labors, an increase in the unemployment rate, and major companies' bankruptcies. However, returning to normal business operations should be done with a safety focus and not be at the cost of global health and wellbeing. Immunity against COVID-19 is going to be a major determinant for a future safe work environment and will reduce the viral infection risk. Therefore, PI is suggesting that if an employee has antibodies against SARS-CoV-2 confirmed by serological testing, he or she could go back to work safely with taking the necessary precautions.

DETAILED DESCRIPTION:
Coronavirus (SARS-CoV2) appeared first in China late 2019 and caused an acute respiratory disease referred as Coronavirus disease 2019 (covid-19). SARS-CoV2 is considered by the World Health Organization (WHO) as pandemic and affected nations worldwide, leading to close borders and major economical struggle. The ongoing viral threat due to the lack of effective therapies and vaccination might prolonged this economical challenge and many businesses will face huge financial constrains leading to laying off labors, increase in the unemployment rate and major companies' bankruptcies. However, returning to normal business operation should be done with a safety focus and not be at the cost of the global health and wellbeing. Immunity against COVID-19 is going to be a major determinant for future safe work environment and will reduce the viral infection risk. Therefore, PI is suggesting that if an employee has antibodies against SARS-CoV-2 confirmed by serological testing, he or she could go back to work safely with taking the necessary precautions.

Materials and Methods: Oncology medical staffs directly involved with patients will be serologically tested using the SARS-CoV-2 IgG assay kit (Abbott Diagnostics, US). If Participants were IgG positive, partcipants will be assumed as immune and therefore, could join the work forces. If partcipants tested negative, partcipants will undergo molecular testing using the RealStar® SARS-CoV-2 RT-PCR Kit RUO (Altona Diagnostics, Germany) to confirm freedom from COVID-19 and then partcipants could join as safe work environment. However, if Positive PCR, partcipants will be quarantined for 14 days or until 2 negative PCR obtained as per the standard Saudi Ministry of Health (MOH) guidelines.

Conclusion: by confirming that healthcare providers have antibodies against SARS-CoV-2 virus and/or their respiratory samples prove the absence of the virus, they can be considered safe and can report to work. By doing so, PI could facilitate going back to normal life and ultimately help improving healthcare functionality as well as overall businesses operation.

ELIGIBILITY:
Inclusion Criteria:

* all Health care provider at KFSH D

Exclusion Criteria:

* NA

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-05-17 (Estimated); Primary Completion 2020-11-16 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Health care provider safe return to work | two weeks from giving serum or swab sample
  by confirming that healthcare providers have antibodies against SARS-CoV-2 virus and/or their respiratory samples prove the absence of the virus, they can be considered safe and can report to work. By doing so, we could facilitate going back to normal life and ultimately help improving healthcare functionality as well as overall businesses operation.

CONTACTS AND LOCATIONS:
Locations (1):
- king Fahad specialist hospital, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No